CLINICAL TRIAL: NCT00598091
Title: A Phase I Study of the Combination of Gemcitabine Plus Dasatinib in Patients With Refractory Solid Tumors With an Expanded Cohort in Advanced Pancreatic Cancer
Brief Title: A Phase I/Expansion Study of Dasatinib
Acronym: Gem/Dsat
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low accrual, unable to meet endpoint in timely manner
Sponsor: Duke University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pro00012976; 9335 (Other: Duke legacy protocol number)
Record Dates: First submitted 2007-12-26; First posted 2008-01-18 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2012-11

CONDITIONS: Refractory Solid Tumors; Pancreatic Adenocarcinoma
Keywords: Solid Tumors; Phase I; Expanded Cohort; Pancreatic Cancer; Dasatinib; Gemcitabine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: gemcitabine; Drug: dasatinib
- B (Active Comparator)
  Interventions: Drug: gemcitabine; Drug: dasatinib

INTERVENTIONS:
Drug: gemcitabine — 1000mg/m2, Days 1, 8, 15
  Other Names: Gemzar
  Arms: A
Drug: dasatinib — 50mg, PO, QD
  Other Names: Sprycel
  Arms: A
Drug: gemcitabine — 1000mg/m2, days 1, 8, 15
  Other Names: Gemzar
  Arms: B
Drug: dasatinib — 50mg, PO, BID
  Other Names: Sprycel
  Arms: B

SUMMARY:
The purpose of this study is to find the highest dose of the drugs gemcitabine and dasatinib that can be given for the treatment of pancreatic cancer. Gemcitabine (also called Gemzar™)is a drug that is given intravenously. Dasatinib (also called Sprycel™) is a tablet and will be taken by mouth.

Gemcitabine is approved by the Food and Drug Administration (FDA) for the treatment of advanced breast, lung and pancreatic cancer. Dasatinib is approved by the FDA for the treatment of chronic myeloid leukemia (CML), acute lymphoblastic leukemia or for patients that are resistant to imatinib mesylate (Gleevec™ ).

This study will try to find the highest doses of these drugs that can be tolerated when taken in combination. The study will also look at how the drugs work in the body, and will see if there is any effect on pancreatic cancer.

DETAILED DESCRIPTION:
This open-label, multicenter, non-randomized phase I trial of gemcitabine plus once and twice daily dasatinib is designed to assess the safety, tolerability, maximum tolerated dose/recommended phase II dose, and preliminary efficacy of this combination in adult patients with advanced solid tumors and with previously untreated metastatic pancreatic cancer. Patients will be accrued at Duke University Medical Center, the Duke Oncology Network, the University of North Carolina at Chapel Hill and Wake Forest Baptist Medical Center

Patients will be accrued to either of the gemcitabine/dasatinib arms in alternating sequential order. In the case where there is an open slot on a particular arm but not the alternative, the enrolled patient will be assigned to that open slot. For example, at the start of the trial, patient #1 will be treated on the gemcitabine with dasatinib twice daily dosing arm, patient #2 on the gemcitabine with dasatinib once daily dosing arm, patient #3 on the gemcitabine with dasatinib twice daily dosing arm, and so on. However, if, due to cohort expansion there is a slot available on one treatment arm but not the other, the patient will be accrued to the open slot.

Additionally, if one arm is held, delayed, or not pursued, accrual to the alternate arm may continue. Patients and their treating physicians will not be able to choose on their own which treatment arm that patient will be assigned to. This enrollment procedure will be the procedure for the entire trial.

For the dose escalation portion of the trial, patients will only be accrued at Duke University Medical Center. For the expanded cohort portion of patients with previously untreated metastatic pancreatic cancer treated at the recommended phase II dose of each arm, patients may be accrued at Duke University Medical Center,and the sites listed above.

NOTE: The first stage closed as of December 2008. Subjects will only be enrolled into the second stage of the this study.

* Toxicity will be assessed every visit, and as clinically indicated.
* Dose limiting toxicities will be assessed during cycle 1.
* Efficacy will be assessed every 2 cycles, and as clinically indicated.
* Plasma biomarkers will be assessed at baseline and at every restaging.
* Tissue based biomarkers (tumor and granulation tissue) will be assessed in up to 15 patients treated at Duke only. Tissue biopsy sets (a 4mm "stimulus" biopsy and a 5mm "granulation" tissue biopsy, both in the same location) will also be done both pre-treatment and on-treatment. Pre-treatment biopsies will be done on days -7 and 1, respectively. On-treatment biopsies will be done on days 1 and 8, respectively.

ELIGIBILITY:
Inclusion Criteria:

Eligibility Criteria Specific for Dose Escalation Phase

* Patients must have histologically confirmed solid tumor malignancy that is metastatic or unresectable and for which standard therapy would include gemcitabine or for which standard curative or palliative measures do not exist or are no longer effective.
* Patients must not have had radiation therapy, hormonal therapy, biologic therapy or chemotherapy for cancer within the 28 days prior to study day 1.

Eligibly Criteria Specific for Expansion Phase at Recommended Phase II Dose

* Histologically or cytologically documented adenocarcinoma of the pancreas.
* Metastatic pancreatic cancer as documented by radiologic study or surgical evidence of metastatic disease.
* No prior chemotherapy for metastatic pancreatic disease. Patients may have received a radiosensiting dose of 5-fluorouracil or capecitabine or other agents used as radiosensitizers with concurrent radiation therapy.
* Last dose of adjuvant chemotherapy must be at least 4 weeks prior to day 1 of the study drug treatment
* Prior radiation therapy is allowed. prior to day 1 of the study drug treatment. At least 4 weeks must have elapsed to baseline or grade 1.
* No prior treatment with gemcitabine or dasatinib in the adjuvant or metastatic setting.
* Prior gemcitabine only allowed if the gemcitabine was administered in the adjuvant setting and > 6 months has elapsed between diagnosis of metastatic disease and last gemcitabine treatment.
* No history for other carcinomas within the last five years, except cured non-melanoma skin cancer, curatively treated in-situ cervical cancer, or localized prostate cancer with a current PSA of <1.0 mg/dL on 2 successive evaluations, at least 3 months apart, with the most recent evaluation no more than 4 weeks prior to day 1 of the study drug treatment. .

Eligibility Criteria for All Subjects

* Age >18 years.
* Karnofsky performance status >70%.
* Life expectancy of at least 3 months.
* Ability to understand and the willingness to sign a written informed consent document.
* Must meet lab requirements as defined in the protocol
* Patients should be capable of taking oral medications for prolonged compliance.
* Sexually active women of childbearing potential must use an effective method of birth control.
* All WOCBP MUST have a negative pregnancy test within 7 days prior to first receiving investigational product.
* Pregnant and/or lactating women will be excluded from this study.

Exclusion Criteria:

* Patients who have had radiation therapy, hormonal therapy, biologic therapy, or chemotherapy for cancer within 28 days prior to day 1 of the study drug treatment. Patients receiving hormonal therapy for metastatic prostate or breast cancer may continue hormonal therapy.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to day 1 of the study drug treatment
* Core biopsy or other minor surgical procedure excluding study-related procedures or placement of a vascular access device within 7 days prior to expected start of treatment.
* Patients who have received any other investigational agents within the 28 days prior to day 1 of the study drug treatment.
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter drug absorption
* History of myocardial infarction, unstable angina, cardiac or other vascular stenting, angioplasty, or surgery within 6 months prior to day 1 of the study drug treatment.
* History of stroke or transient ischemic attack within 6 months prior to day of the study drug treatment.
* Uncontrolled congestive heart failure defined as New York Heart Association (NYHA) class II or greater
* Known cardiomyopathy with decreased ejection fraction (less than institutional normal limits)
* Diagnosed or congenital long QT syndrome
* Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes)
* Prolonged QTc interval on pre-study electrocardiogram (> 450 msec)
* Patients with a history of significant bleeding episodes (e.g., hemoptysis, upper or lower GI bleeding) within the previous 6 months of day 1 of the study drug treatment
* Evidence of bleeding diathesis or coagulopathy. Patients on therapeutic anticoagulation may be enrolled provided that they have been clinically stable on anti-coagulation for at least 2 weeks prior to day 1 of the study drug treatment
* History of significant bleeding disorder unrelated to cancer
* Medications that inhibit platelet function
* Fluid retention (i.e. pleural effusion, ascites, edema) grade > 2.
* A known history of HIV seropositivity, hepatitis C virus, acute or chronic active hepatitis B infection, or other serious chronic infection requiring ongoing treatment.
* Patients currently taking drugs that are generally accepted to have a risk of causing Torsades de Pointes
* Patients actively taking inhibitors or inducers of CYP3A4
* Patients actively taking proton pump inhibitors or H2 antagonists
* Other concurrent severe and/or poorly controlled medical condition that could compromise safety of treatment
* Any psychiatric illness/social situations that would limit safety or compliance with study requirements or may interfere with the interpretation of the results.
* Patients unwilling to or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-04; Primary Completion 2010-06 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
To determine the MTD/Recommended Phase II Dose (RPTD) of gemcitabine plus dasatinib once daily and twice daily dosing in patients with advanced solid tumors | Phase I portion of the study

SECONDARY OUTCOMES:
To describe any dose limiting toxicities for these regimens | Every 28 days or as clinically indicated
To describe and non-dose limiting toxicities for these regimens | Every 28 days or as clinically indicated
To preliminarily describe markers of efficacy for gemcitabine plus dasatinib in patients with previously untreated metastatic pancreatic cancer: response rate, progression free survival, overall survival. | Every 8 weeks
To preliminarily describe changes in blood and urine based biomarkers,at baseline compared to first restaging and at progression, for patients with previously untreated metastatic pancreatic cancer treated on the expanded cohorts at the MTD/RPTD. | baseline, first restaging, progression

CONTACTS AND LOCATIONS:
Overall Officials: Hope C Uronis, MD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - UNC Lineberger, Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina